CLINICAL TRIAL: NCT06267612
Title: Long-term Follow-up Study of Corheart 6 Left Ventricular Assist System as Treatment of Patients With Advanced Heart Failure
Brief Title: Corheart 6 LVAS Long-term Follow-up Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Zhibing Qiu, Professor, Nanjing First Hospital, Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20231109-11
Record Dates: First submitted 2024-02-02; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Corheart 6 LVAS (Experimental): Corheart 6 Left Ventricular Assist System (Corheart 6 LVAS) to be used on patients with advanced heart failure.
  Interventions: Device: Corheart 6 Left Ventricular Assist System

INTERVENTIONS:
Device: Corheart 6 Left Ventricular Assist System — Implantation of left ventricular assist device for hemodynamic support

SUMMARY:
The purpose of this clinical study is to explore the long-term efficacy and safety of the Corheart 6 Left Ventricular Assist System (LVAS) as a treatment for patients with advanced heart failure.

The study will be a single-arm, prospective, single-center, non-blinded, and non-randomized study with a follow-up duration of five years.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 18 years.
* 2. The patient or legal representative is willing to participate in the study and offers informed consent.
* 3. Body surface area (BSA) ≥ 1.0 m^2.
* 4. Females of childbearing age must agree to use adequate contraception.
* 5. Patients with NYHA Class IV heart failure symptoms who have failed to be reversed by standardized treatment with oral anti-heart failure drugs.
* 6. Left Ventricular Ejection Fraction (LVEF) ≤ 35%, and at least one of the following conditions occurs:
* a. Fail to be reversed by or be weaned from intra-aortic balloon pump (IABP), extracorporeal membrane oxygenator (ECMO), or other short-term mechanical circulatory support.
* b. Rely on continuous intravenous administration of one or more vasoactive or inotropic drugs.
* c. Meeting the diagnostic criteria of cardiogenic shock: blood pressure < 90/60mmHg, cardiac index < 2.0 L/min/m^2 (optional), and pulmonary capillary wedge pressure > 18mmHg (optional).

Exclusion Criteria:

* 1. Etiology of heart failure due to or associated with uncorrected thyroid disease, obstructive hypertrophic cardiomyopathy, or pericardial disease.
* 2. Presence of an active, uncontrolled infection confirmed by a combination of clinical symptoms and laboratory tests.
* 3. Technical obstacles which pose an inordinately high surgical risk, in the judgment of the investigator.
* 4. Intolerance to anticoagulant or antiplatelet therapies or any other peri/postoperative therapy the investigator will require based on the patient's health status.
* 5. Patients require bi-ventricular assist device support.
* 6. Pregnancy.
* 7. Presence of moderate to severe aortic insufficiency or a history of the mechanical aortic valve that will not be converted to a bioprosthesis or oversewn at the time of implantation.
* 8. History of any organ transplantation.
* 9. Presence of uncorrected thrombocytopenia or severe coagulopathy, such as diffuse intravascular coagulation.
* 10. TBIL (total bilirubin) > 3.0 mg/dL within 48 hours prior to implantation.
* 11. Serum creatinine (SCr) > 3.0 mg/dL within 48 hours prior to implantation or may require dialysis.
* 12. Presence of severe chronic obstructive pulmonary disease (COPD) or restrictive lung disease or a diagnosis of primary pulmonary hypertension.
* 13. Presence of pulmonary embolism within 3 weeks prior to implantation.
* 14. Pulmonary artery systolic pressure exceeds 60mmHg, combined with at least one of the following 2 parameters demonstrating that pulmonary vascular resistance did not respond to drug therapy:
* a. Pulmonary vascular resistance greater than 8 wood units.
* b. The transpulmonary differential pressure exceeds 20mmHg.
* 15. Established and untreated abdominal or thoracic aortic aneurysm > 5cm in diameter.
* 16. Presence of severe peripheral vascular disease with resting pain or extremity ulceration.
* 17. Psychiatric disease/disorder, irreversible cognitive dysfunction or psychosocial issues that are likely to impair compliance with the study protocol and LVAS management, or brain death from various causes.
* 18. History of documented disabling stroke within 90 days prior to implantation, a history of cerebrovascular disease, or the presence of uncorrected severe bilateral carotid artery stenosis.
* 19. History of acute myocardial infarction within 60 days prior to implantation, judged by the investigator to have a risk of myocardial rupture or other surgical high-risk difficult-to-control bleeding, etc.
* 20. Expected lifetime of less than 1 year due to malignant tumor or other disease.
* 21. Participation in any other clinical study that may influence the results of this study.
* 22. Other circumstances that are unforeseen and determined by the researcher to be unsuitable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-10 (Estimated); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Device implantaion success rate at 24 months post-implantation | Up to 24 months post-implantation
  Device implantation success is defined as:
  * A. Electively transplanted or explanted prior to 24 months or
  * B. Alive at 24 months, and
  * I. Have not experienced a stroke with a modified Rankin Score > 3, and
  * II. Have not received a device replacement or exchange due to a device malfunction, and
  * III. Have not received an urgent transplant due to a device malfunction.

SECONDARY OUTCOMES:
Quality of Life as measured by the Kansas City Cardiomyopathy Questionnaire-23 (KCCQ-23) | Baseline, at 6 months, 12 months, 18 months, and 24 months post-implantation
  Scores range from 0 to 100. Higher scores indicate better quality of life and fewer heart failure symptoms.
Quality of Life as measured by the EuroQoL-5D-5L (EQ-5D-5L) questionnaire | Baseline, at 6 months, 12 months, 18 months, and 24 months post-implantation
  The scores from the 5 dimensions are summed for the total score, with higher scores indicating more problems and a worse quality of life.
Functional status as measured by the Six Minute Walk Test (6MWT) | Baseline, at 6 months, 12 months, 18 months, and 24 months post-implantation
  The more meters a patient can walk over baseline indicates improvement in functional status.
Functional status as measured by the New York Heart Association (NYHA) Classification | Baseline, at 6 months, 12 months, 18 months, and 24 months post-implantation
  NYHA class categorizes patients by the severity of their heart failure symptoms. As the class increases, the degree of symptoms is more severe indicating worse functional status.
Stroke severity as assessed with the National Institutes of Health Stroke Scale (NIHSS) score | Baseline, at 6 months, 12 months, 18 months, and 24 months post-implantation, and as a stoke event occurs, from baseline to 24 months post-implantation
  Scores range from 0 to 42. Higher scores indicate more severe disability
Stroke severity as assessed by the modified Rankin Scale (mRS) score | Baseline, at 6 months, 12 months, 18 months, and 24 months post-implantation, and as a stoke event occurs, from baseline to 24 months post-implantation
  Scores range from 0 to 6. Higher scores indicate more severe disability
Adverse events | As they occur, from baseline to 24 months post-implantaion
  Frequency and incidence of all anticipated adverse events
Device-related re-operations | As they occur, from baseline to 24 months post-implantaion
  Frequency and incidence of all device-related re-operations
Device-related re-hospitalizations | As they occur, from initial hospital discharge to 24 months post-implantation
  Frequency and incidence of all device-related re-hospitalizations
Overall survival | Up to 60 months post-implantation
  Overall survival at 60 months post-implantation

CONTACTS AND LOCATIONS:
Overall Officials: Zhibing Qiu, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No